CLINICAL TRIAL: NCT06981247
Title: m-Lifestyle Intervention for Employees (m-LIfE): Protocol for a Pilot Cluster Randomized Controlled Trial on Cardiovascular Disease Prevention Strategies
Brief Title: Cardiovascular Disease Prevention Strategies for High-risk Urban Sedentary Employees in Karachi, Pakistan
Acronym: m-LIfE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Aysha Almas, Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ERC No. 2025-9680-29143; 5D43TW011625 (NIH)
Record Dates: First submitted 2025-04-19; First posted 2025-05-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-05

CONDITIONS: Physical Activity; Life Style; Dietary Habits; Cardiovascular Diseases
Keywords: Primary care; Cardiology; Preventive medicine; risk perception; cardiovascular health; CVD; Sedentary lifestyle; mHealth; Digital health; Feasibility
MeSH Terms: conditions — Motor Activity; Feeding Behavior; Cardiovascular Diseases; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- m-LIfE (Experimental): Participants in the intervention arm will receive mHealth application (m-LIfE). The application will be installed on participants' personal mobile phones, and each participant will be provided with a unique user ID and password.
  Interventions: Behavioral: m-LIfE: mobile based lifestyle intervention for employees to increase their physical activity and promote healthy diet.
- Routine care arm (Other): Participants in the routine care arm will receive basic educational material in the form of paper-based pamphlets without any active intervention by the study team.
  Interventions: Other: Routine care arm

INTERVENTIONS:
Behavioral: m-LIfE: mobile based lifestyle intervention for employees to increase their physical activity and promote healthy diet. — The m-LIfE will primarily deliver healthy lifestyle educational content, provide customized strategies for PA, and offer participants the option to enter their daily intake of fruits and vegetables through Food Log feature. m-LIfE will track PA and diet, send tailored reminders, and provide motivational messages. Participants will receive two text messages daily: a goal reminder in the morning and feedback or reflection on their progress in the evening. Additionally, they will receive one motivational message at the end of each week to sustain their motivation. Personalized feedback will also be provided through the application, featuring graphs to illustrate daily, weekly, and monthly progress.
  To support participants further, the application will enable two-way communication, allowing users to seek assistance and ask questions from the research team. A dedicated contact number will be made available within the app to facilitate direct communication.
  Arms: m-LIfE
Other: Routine care arm — Participants in the routine care arm will receive educational material in the form of paper-based pamphlets to ensure they still benefit from basic health information on CVD risk prevention. They will continue their usual work routines without access to the app, but their PA and dietary habits will be assessed at baseline, post-intervention and at follow-up for comparative purposes.
  Arms: Routine care arm

SUMMARY:
Heart diseases and other non-communicable diseases are serious health issues in countries like Pakistan. Many people who work in offices, like bank employees, sit for more than 8 hours a day. This is called a sedentary lifestyle, and it increases the risk of heart diseases.

This research project aims to find out if a newly developed context specific mobile phone application can help these sedentary employees to improve their lifestyle. The app, called m-LIfE (mHealth-based Lifestyle Intervention for Employees), will be designed to help employees to move more during the day and eat healthier food like fruits and vegetables.

The study will involve bank employees in urban Karachi, Pakistan. They will be divided into two arms:

Intervention arm: Participants in this arm will use the m-LIfE app for 12 weeks. They will get reminders and tips to take breaks, exercise, and eat healthy.

Routine care arm: Participants in this arm will receive printed basic educational material about prevention of risk factors of heart diseases and improving lifestyle.

After the 12 weeks of intervention, there will be a follow-up period at 4th week to check if participants are maintaining healthy habits.

This study could help find simple and affordable ways to improve the health of office workers and reduce pressure on the healthcare system.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) are the leading cause of mortality globally, with developing countries bearing a disproportionate burden of associated risk factors. Alarmingly, the age of onset of CVD is decreasing in these settings. Despite the significant burden, preventive strategies targeting modifiable risk factors often receive insufficient attention. Pakistan, as the fifth most populous country in the world and a low and middle-income country (LMIC) with a fragile healthcare system, relies heavily on out-of-pocket payments for healthcare (73% of the population). In this context, addressing CVD risk factors at the population level and targeting high-risk populations becomes an essential strategy for combating CVD.

The banking sector in particular has been facing a tremendous change for several years due to the increasing number of new entrants, which has increased competition among the banks. Economic uncertainties and political instability have also affected the industry and consequently the health outcomes of its employees who are considered high risk urban sedentary workers as they spend more than 8 hours of their daytime sitting with minimal physical activity (PA) and consuming high lipid diet. This behavior predisposes them to CVD unless they take preventive health behaviors (engage in regular PA, increase fruit and vegetable intake, and reduce fatty meals, sugar, and salt intake). Lifestyle modification aimed at improving PA and dietary habits is the first-line approach to reducing cardiovascular risk. However, the feasibility of implementing such strategies in urban environments needs to be examined. Currently, little is known about which intervention components would be most effective in improving the lifestyle behaviors of bank employees.

Pertinently, the workspaces of most bank branches in Pakistan lack suitable areas for relaxation or PA, further exacerbating the sedentary nature of their work. Consequently, this high-risk group requires targeted efforts to increase their knowledge and address their lifestyle behaviors for effective CVD prevention. Therefore, the development and testing of strategies specifically tailored to this occupational group are of utmost importance.

The overall aim of this research project is to develop and assess the feasibility of m-LIfE (mHealth-based Lifestyle Intervention for Employees) to improve lifestyle in high-risk urban sedentary employees (bank employees) from Karachi, Pakistan. The specific objectives are (1) To explore awareness (perception and preferences) about CVD and its prevention among high-risk sedentary employees, and design m-LIfE (2) To assess feasibility of m-LIfE versus routine care among high-risk sedentary employees. The secondary objective is to report potential efficacy on lifestyle (PA and dietary intake) in both m-LIfE and routine arm.

This study will employ a mixed-methods approach, beginning with an exploratory qualitative phase and followed by a pilot cluster randomized controlled trial (cRCT). The qualitative component will explore awareness, perceptions, and preferences regarding CVD and its prevention. Following this, m-LIfE app will be developed using human centered design approach.

The pilot cRCT will evaluate the feasibility and potential efficacy of the m-LIfE over a 12-week intervention period, with a 4-week follow-up. Eight clusters (bank branches) will be randomly selected out of 313 branches across Karachi, out of which four will be randomized to the m-LIfE intervention, and four clusters will serve as the routine care arm. The study will be conducted in branches of three commercial banks (one public and two private) located in urban Karachi, Pakistan.

ELIGIBILITY:
Inclusion Criteria:

• At least 6 months of job experience in any bank

Exclusion Criteria:

* Diagnosed case of myocardial infarction, stroke, coronary heart disease, cerebrovascular disease, or peripheral arterial diseases
* Pregnant women
* Individuals with acute illnesses that limit physical activity

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of m-LIfE application (Recruitment Rate) | Recruitment rate will be measured at baseline.
  Recruitment rate will be measured as the percentage of participants enrolled out of the total number of eligible participants invited to receive m-LIfE intervention. The trial will be considered feasible if recruitment rate exceeds 70%.
  Units of Measure: Percentage (%)
Feasibility of m-LIfE application (Retention Rate) | Retention rate will be measured at post-intervention (Week 12, immediately after the intervention ends)
  Retention rate will be measured as the percentage of participants who complete the post-intervention assessment at 12 weeks, out of those who were initially enrolled. The intervention will be considered feasible if the retention rate exceeds 70%.
  Units of Measure: Percentage (%)
Feasibility of m-LIfE application (Treatment Fidelity) | Treatment fidelity will be measured at post-intervention (Week 12, immediately after the intervention ends)
  The treatment fidelity rate will be measured as the percentage of planned health-promoting sessions successfully delivered during the 12-week intervention period.
  The intervention will be considered feasible if the treatment fidelity rate exceeds 70%.
  Units of Measure: Percentage (%)

SECONDARY OUTCOMES:
Potential efficacy of m-LIfE application (Physical activity) | Data will be collected at three time points: baseline (Week 0), post-intervention (Week 12), and follow-up (Week 16, four weeks after the intervention ends).
  The duration of physical activity will be measured as the mean change in the daily step count.
  Unit of Measure: Step count

OTHER OUTCOMES:
Change in waist circumference | Data will be collected at three time points: baseline (Week 0), post-intervention (Week 12), and follow-up (Week 16, four weeks after the intervention ends).
  It will be measured as the mean change in the waist circumference. Unit of Measure: Centimeters (cm)
Change in body mass index | Data will be collected at three time points: baseline (Week 0), post-intervention (Week 12), and follow-up (Week 16, four weeks after the intervention ends).
  It will be measured as the mean change in the body mass index. Unit of Measure: kilograms per meter squared (kg/m²)
Changes in vegetable intake | Data will be collected at three time points: baseline (Week 0), post-intervention (Week 12), and follow-up (Week 16, four weeks after the intervention ends).
  It will be measured as the mean change in the number of servings of vegetables consumed per week by participants.
  Unit of Measure: Servings per week
Changes in fruits intake | Data will be collected at three time points: baseline (Week 0), post-intervention (Week 12), and follow-up (Week 16, four weeks after the intervention ends).
  It will be measured as the mean change in the number of servings of fruits consumed per week by participants.
  Unit of Measure: Servings per week
Change in diastolic blood pressure | Data will be collected at three time points: baseline (Week 0), post-intervention (Week 12), and follow-up (Week 16, four weeks after the intervention ends).
  It will be measured as the mean change in the Diastolic blood pressure reading. Unit of Measure: Millimeters of mercury (mmHg)
Change in systolic blood pressure | Data will be collected at three time points: baseline (Week 0), post-intervention (Week 12), and follow-up (Week 16, four weeks after the intervention ends).
  It will be measured as the mean change in the systolic blood pressure reading. Unit of Measure: Millimeters of mercury (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Aysha Almas, PhD, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
We plan to share deidentified IPD with other researchers. The shared data will include deidentified participant behavioral risk factors, and other relevant variables collected during the study. Access to the data will be granted upon reasonable request. A data-sharing agreement that outlines the intended use of the data will be signed. Researchers requesting the data will need to adhere to ethical guidelines and data protection policies.
Supporting Information: Study Protocol
Time Frame: Soon after the publication of trial with no end date
Access Criteria: Researchers will need to submit a formal request to the PI, explaining the purpose of their request and how they plan to use the data. Access will be granted primarily for the purpose of verifying the results presented in the study. Any secondary analyses or additional studies using the IPD will require explicit permission from the PI.

REFERENCES:
- [Background] Elahi A, Ali AA, Khan AH, Samad Z, Shahab H, Aziz N, Almas A. Challenges of managing hypertension in Pakistan - a review. Clin Hypertens. 2023 Jun 15;29(1):17. doi: 10.1186/s40885-023-00245-6. PMID 37316940
- See also: This URL links to the World Health Organization website, which provides the latest facts about cardiovascular disease (CVD) and its risk factors. — https://www.who.int/news-room/fact-sheets/detail/cardiovascular-diseases-(cvds)